CLINICAL TRIAL: NCT00759928
Title: Pharmacokinetic Trial of Sorafenib and Erlotinib in Patients With Refractory Solid Tumors
Brief Title: PK Trial of Sorafenib & Erlotinib in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 175
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Refractory Solid Tumors
Keywords: Refractory Solid Tumors; Unresectable Stage III/IV; Sorafenib; Erlotinib; Pharmacokinetics
MeSH Terms: interventions — Erlotinib Hydrochloride; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib/Sorafenib (Experimental): Patients will receive erlotinib 150 mg once daily by mouth and sorafenib 400 mg twice daily by mouth. The study will begin with a 2-week run-in period (which will begin on Day 14 of the study, and continue through Day 1 of the study), in which erlotinib will be dosed alone at 150 mg once daily. Patients will continue taking erlotinib as a single agent at 150 mg once daily through Day 1. After the 2-week run-in period, patients will receive continuous dosing of both agents (erlotinib 150 mg once daily and sorafenib 400 mg twice daily) in cycles of 28 days each. Toxicity will be assessed every cycle (every 4 weeks) for all patients. Because this is not an efficacy study, restaging tumor measurements will be at the discretion of the physician every 8 weeks during treatment. Patients with objective response or stable disease will continue therapy; patients with disease progression or unacceptable toxicity will be discontinued from the study.
  Interventions: Drug: Erlotinib; Drug: Sorafenib

INTERVENTIONS:
Drug: Erlotinib — 150 mg once daily by mouth
  Other Names: Tarceva
Drug: Sorafenib — 400 mg twice daily by mouth
  Other Names: Nexavar

SUMMARY:
Two cohorts of patients will be enrolled: Cohort A will consist of patients who are current smokers, and Cohort B will consist of patients who are current nonsmokers. There will be 24 patients enrolled in each cohort. Nonsmokers are patients who have not consumed tobacco or nicotine-containing products for 1 year before the start of the study. Patients classified as current smokers must have smoked a minimum of 10 cigarettes per day for up to 1 year. Patients who have smoked 1-9 cigarettes per day for up to 1 year, or more than 10 cigarettes per day for less than 1 year will not be eligible for this study.

DETAILED DESCRIPTION:
Compared with supportive care alone, erlotinib has been associated with improved overall survival in patients with Refractory Solid Tumors; however, this absolute benefit is limited for the majority of patients. Incorporating other biologic agents into the second- or third-line treatment setting may prove to be a successful strategy in improving treatment efficacy (which has been recently demonstrated in several tumor types). Additionally, recent data suggest that smoking may influence the pharmacokinetic (PK) profile of erlotinib by increasing the metabolic clearance. Data suggest that the geometric mean erlotinib AUC(0-inf) and C(24h) are significantly decreased in smokers compared with nonsmokers (Hamilton et al. 2006). For this reason, this trial will enroll separate cohorts of patients who are current smokers and patients who are nonsmokers. Nonsmokers are patients who have not consumed tobacco or nicotine-containing products for 1 year before the start of the study. Patients classified as current smokers must have smoked a minimum of 10 cigarettes per day for up to 1 year.

ELIGIBILITY:
1. Histologically confirmed incurable solid tumors refractory to standard treatment or for which there is no known standard treatment.
2. Two cohorts of patients will be enrolled: Cohort A will consist of patients who are current smokers, and Cohort B will consist of patients who are current nonsmokers. Nonsmokers are patients who have not consumed tobacco or nicotine-containing products for 1 year before the start of the study. Patients classified as current smokers must have smoked a minimum of 10 cigarettes per day for <1 year.
3. Patients must have evaluable disease.
4. Recovery from any toxic effects of prior therapy to grade 1 per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
5. Completion of radiation therapy at least 21 days prior to the start of study treatment (not including palliative local radiation).
6. An Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Absolute neutrophil count (ANC) >1,500/mL and platelets >75,000/mL (within 7 days prior to study treatment).
8. Hemoglobin >9 g/dL (within 7 days prior to treatment). Patients may be transfused or receive erythropoietin to maintain or exceed this level where otherwise indicated.
9. International normalized ratio (INR) <1.5 or prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits (WNL) of the institution (if patient is not on anti-coagulation therapy; patients receiving anticoagulation treatment with an agent such as warfarin or heparin may be allowed to participate with the therapeutic range established prior to the initiation of study treatment).
10. Serum creatinine <1.5 x the institutional upper limit of normal (ULN) within 7 days prior to study treatment. If the absolute value is greater than 2 mg/dL, the creatinine clearance (calculated according to the Cockcroft-Gault formula) must be > 45 mL/min for the patient to be eligible for the study.
11. Transaminases <3 x the institutional ULN (except if there is known hepatic metastasis, wherein transaminases may be <5 x institutional ULN).
12. Total bilirubin <1.5 times ULN.
13. Patients must be able to understand the nature of this study, give written informed consent, and comply with study requirements.
14. Agreement of female patients of childbearing potential and male patients who have partners of childbearing potential to use an effective form of contraception to prevent pregnancy during treatment, and for a minimum of 90 days thereafter. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.

Exclusion

1. Patients with untreated brain metastases. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis. Patients who have a history of brain metastases that has been treated by surgery or radiation therapy > 4 weeks with no signs of Central Nervous System (CNS) progression are allowed.
2. Women who are pregnant or lactating.
3. Patients whose last dose of chemotherapy, immunotherapy, or investigational drug therapy was completed < 21 days prior to receiving study drug
4. Significant cardiac disease within 90 days of starting study treatment including:

   * superior vena cava syndrome;
   * new onset angina;
   * congestive heart failure (CHF) > Class 2 per New York Heart Association (NYHA) classification (see Appendix B);
   * ventricular arrhythmia;
   * valvular heart disease.
5. Myocardial infarction (MI) within 6 months prior to initiation of study treatment.
6. Cardiomegaly on chest imaging or CHF > Class 2 per NYHA classification (see Appendix B) unless the left ventricular ejection fraction (LVEF) is within normal range for the institution within 3 months of initiating therapy.
7. Poorly controlled hypertension (defined as systolic blood pressure [BP] >150 mmHg and/or diastolic blood pressure >90 mmHg on anti-hypertensive medications).
8. Unstable angina (anginal symptoms at rest).
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
10. Presence of cardiac disease that, in the opinion of the investigator, increases the risk of ventricular arrhythmia.
11. A serious active infection (> grade 2) at the time of treatment
12. A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
13. A major surgical procedure within 28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study.
14. Any minor surgery must be completed within 7 days prior to beginning study treatment.
15. Use of rifampin, St. John's wort, or other potent inducers of CYP3A4 are not permitted from Day -14 through Day 15 of the study (see Appendix C).
16. Use of ketoconazole and other potent inhibitors of CYP3A4 are not permitted from Day -14 through Day 15 of the study (see Appendix C).
17. Stroke or transient ischemic attack (TIA) within the past 6 months.
18. Any prior history of hypertensive crisis or hypertensive encephalopathy.
19. Pulmonary hemorrhage/bleeding event > grade 2 within 28 days of study treatment.
20. Any other non-pulmonary hemorrhage/bleeding event> grade 3 within 28 days of study treatment.
21. Evidence or history of bleeding diathesis or coagulopathy.
22. Serious non-healing wound, ulcer, or bone fracture.
23. Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.
24. Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease.
25. Patients who smoke 1-9 cigarettes per day during the year before study entry or patients who have smoked for <1 year will not be eligible for this study.
26. Any condition that impairs the patient's ability to swallow whole pills.
27. Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetics (PK) of erlotinib when administered in combination with sorafenib on a continuous schedule in Refractory Solid Tumors in patients who are smokers and in patients who are nonsmokers. | 3 months

SECONDARY OUTCOMES:
To evaluate safety of this combination in patients with Refractory Solid Tumors. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Tennessee Oncology, Nashville, Tennessee